CLINICAL TRIAL: NCT02312947
Title: Coblation Versus Cold Adenoidectomy -Safety and Efficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0047-14-HYMC
Record Dates: First submitted 2014-12-06; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- coblation (Active Comparator): coblation adenoidectomy
  Interventions: Device: coblation (COBLATION II surgery system ,CE8001-01)
- cold dissection (Active Comparator): cold dissection adenoidectomy
  Interventions: Device: cold dissection adenoidectomy

INTERVENTIONS:
Device: coblation (COBLATION II surgery system ,CE8001-01) — comparison of two methods of operation : coblation and cold dissection
  Other Names: COBLATION II surgery system ,CE8001-01
  Arms: coblation
Device: cold dissection adenoidectomy — comparison of two methods of operation : coblation and cold dissectionby currete
  Other Names: currete adenoidectomy
  Arms: cold dissection

SUMMARY:
Comparative two methods of adenoidectomy means the coblation adenoidectomy with the cold dissection adenoidectomy specifically inquire which method is safer and more efficient.

DETAILED DESCRIPTION:
Obstructive sleep apnea(osa) in children is a very bother and frequent problem with clinical and behavioral impacts. The hypertrophied adenoid tissue obstructs the air way in the nasopharynx that initiates the common symptoms. The treatment from that concerning problems is in the operation rooms by diversity surgical methods, the very older one is the cold dissection adenoidectomy.

Recently many surgeons use the coblation system as a preferred method for adenoidectomy. This method was proof as a safe and efficient especially referring to the bleeding and the dehydration risk .

Many children that operated by the cold dissection forced to perform another one or two operations presumably due to the adenoid tissue that did not removed completely from the first operation .

our hypothesis is that the coblation systemis a safe and eficient method for adenoidectomy.

The aims of this project is to verify if our theory is corect by blinded comparision between two methods.

ELIGIBILITY:
Inclusion Criteria:

* children with obstructive symptoms
* the children must perform nasopharyngoscopy with clear evidence of obstructive symptoms ( video or polysomnography more than 5 RDI)

Exclusion Criteria:

* without any recent upper respiratory tract infection or clinical suspicious of adenoiditis.
* tonsillectomy
* Non randomalization, not blinded

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-12; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
safety (bleeding , dehydration or any other complications) | percent of bleeding and dehydration
  measure the event of bleeding , dehydration or any other complications

SECONDARY OUTCOMES:
efficacy (pain post operation by scales evaluation) | pain and examination for residual adenoid tissue
  pain post operation by scales evaluation and determination whether adenoid tissue left behind after each methods of operation